CLINICAL TRIAL: NCT04163094
Title: Ovarian Cancer Treatment With a Liposome Formulated mRNA Vaccine in Combination With (Neo-)Adjuvant Chemotherapy
Acronym: OLIVIA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Despite the extension of the original recruitment period, the target number of evaluable patients defined in the study protocol could not be reached and recruitment for the trial was stopped at that point of time.
Sponsor: University Medical Center Groningen (Other)
Collaborators: BioNTech SE (Industry)
Responsible Party: Principal Investigator, Hans W. Nijman, MD PHD, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLIVIA-UMCG-01; 2017-004585-10 (EudraCT Number)
Record Dates: First submitted 2019-11-06; First posted 2019-11-14 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a first-in-human, open label phase I study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Patients will receive 8 W_ova1 vaccinations before and during neoadjuvant chemotherapy and adjuvant chemotherapy.
  Interventions: Drug: W_ova1 Vaccine

INTERVENTIONS:
Drug: W_ova1 Vaccine — Patients will be treated with a W_ova1 vaccine that includes 3 OC TAA RNA-LPX products.

SUMMARY:
This is a first-in-human, open label phase I study in ovarian cancer patients with primary disease eligible for standard-of-care treatment with neo-adjuvant chemotherapy, i.e. 3 cycles carboplatin/paclitaxel, interval surgery and 3 additional cycles carboplatin/paclitaxel. Eight doses of the W_ova1 vaccine will be administered prior and in combination with the (neo-)adjuvant chemotherapy to induce an anti-tumor immune response. Systemic immune responses are determined using peripheral blood mononuclear cells collected before, during and after vaccinations. Intratumoral accumulation of T-cells recognizing vaccine-encoded TAAs will be determined before vaccination in a tumor biopsy and after the 3 cycles of chemotherapy and the 5th vaccination using tumor tissue derived from interval surgery. [18F]FB-IL2 PET-CT will be used for the non-invasive assessment of T-cell activation and correlated to immunohistochemistry tumor tissue data from pre-treatment biopsy and interval debulking surgery

DETAILED DESCRIPTION:
This is a first-in-human, open label phase I intra-patient dose escalation study (vaccination 1 and 2) in OC patients with primary disease eligible for SoC treatment with neo-adjuvant chemotherapy, i.e. 3 cycles carboplatin/paclitaxel, interval surgery and 3 additional cycles carboplatin/paclitaxel.

OC patients will be vaccinated prior and during (neo)-adjuvant chemotherapy with the W_ova1 vaccine, which includes 3 OC TAA RNAs. Vaccines will be administered by means of intravenous injection. A total of eight vaccinations will be administered with intra-patient dose escalation planned for the first two doses, i.e. the first vaccine will contain 50 µg total RNA and the subsequent seven vaccines will contain the target dose of 100 µg total RNA. Dose reductions/modifications to 50, 25 and 14.4 µg are allowed per protocol.

The first two vaccinations will be administered before the start of neo-adjuvant chemotherapy with 7 day time lag (+/- 2 days) between each vaccination. The subsequent 6 vaccinations are scheduled 15 days (+/- 3 days) after the start of each cycle of chemotherapy to avoid overlap with immune-suppressive corticosteroid premedication as well as with the direct effects of the chemotherapy. Patient evaluation will be performed before, during and after vaccination, including history, physical examination, ECOG performance status and toxicity scoring using NCI CTCAE 5.0 toxicity grades. Blood sample collection for bio monitoring by means of a vena puncture will occur before each vaccination. During the two-step dose escalation blood samples will also be collected 6 hours and 24 hours after vaccination. Blood samples will be analyzed for biochemistry, hematology and tumor marker CA-125.

To determine the systemic immune response (primary objective), PBMCs are obtained by venous blood collection at baseline (100 mL) and twice during study related treatment period (60 mL). In addition, three leukaphereses (or 100 mL blood draw alternatively) and four blood draws for ctDNA analysis are scheduled during the trial for each patient.

To determine the intratumoral immune response (secondary objective), tumor material will be collected before vaccination by an image-guided biopsy and during surgery (standard treatment).

The first [18F]FB-IL2 PET-CT (exploratory objective) will occur at baseline and the second [18F]FB-IL2 PET-CT as close to the surgery as possible. These study procedures are optional and patients can still participate in the trial without the [18F]FB-IL2 PET-CT.

In case of premature drop-out, patients will be asked to undergo the leukapheresis (or 100 mL blood draw alternatively) and if possible / feasible, additional tumor material sampling at time of the planned interval surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary epithelial OC patients with measurable tumor lesions (determined by CT or MRI), who are intended to be treated with neo-adjuvant chemotherapy (carboplatin/paclitaxel), subsequent surgery and adjuvant chemotherapy
* Age ≥ 18 years
* Signed informed consent in accordance with institutional and regulatory guidelines
* Adequate access of the tumor for image-guided biopsy
* Adequate (according to the institutional standards) hematology, liver and kidney function to undergo chemotherapy with carboplatin and paclitaxel
* ECOG-performance status of 0 or 1 at screening
* Current BMI > 18.5 and no weight loss of >5% over the past month. Notably, weight loss due to drainage of ascites is not applicable.

Exclusion Criteria:

* History of a second malignancy except for curatively treated low-stage tumors with a histology that can be differentiated from the epithelial OC type
* History of an autoimmune disease, specifically HAV, HBV, HCV and HIV, or any other systemic intercurrent disease or condition that might affect the immunocompetence of the patient, or treatment with systemic highly immunosuppressive therapy (e.g. transplant recipients or patients who underwent a splenectomy)
* Use of systemic continuous corticosteroid therapy (e.g. prednisone i.v. or p.o. >7.5 mg / day).
* Pregnancy or breast feeding
* Participation in a trial with another investigational drug within 30 days prior to the enrolment in this trial
* Any condition that in the opinion of the investigator could interfere with the conduct of the trial.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline W_ova1 vaccine antigen-specific T cells in the peripheral blood (systemic induction / expansion of W_ova1 vaccine antigen-specific T cells). | A PBMC collection is planned at baseline, before start treatment. A further PBMC collection is scheduled after 5 vaccinations before surgery. The post-vaccination PBMC collections are scheduled at approx. 14 days and 2.5 months after final vaccination.
  Number of patients with de novo or increased systemic immune responses (based on the ELISpot Data Analysis Tool 1.0) in the post-vaccination PBMC sample compared to baseline PBMC sample to at least one of the three vaccine antigens

SECONDARY OUTCOMES:
Change from baseline W_ova1 vaccine antigen-specific T cells in the tumor (Intratumoral induction / expansion of W_ova1 vaccine antigen-specific T cells) | Tumor material is collected at baseline by biopsy and compared to tumor material collected during standard-of-care cytoreductive surgery (mid-vaccination, week 12)
  Number of patients with a significant increase (p<0.05) in CD8-cell density (CD8-cells / mm2 cancer epithelium [cytokeratin-positive area]) in tumor (pre- and post-treatment biopsy)
Progression free survival | Up to 2 years from disease diagnosis
  PFS defined as the number of patients alive without any progress or recurrence (local or regional, or distant) and death due to any cause
Safety and tolerability of repetitive doses of the W_ova1 vaccine in combination with carboplatin/paclitaxel | Up to 28 days after last vaccination
  Number of patients with AEs, and SAEs

OTHER OUTCOMES:
Change from baseline intratumoral visualization of CD25+ T cells using [18F]FB-IL2 PET-CT | Baseline [18F]FB-IL2 PET-CT compared to [18F]FB-IL2 PET-CT before standard of care cytoreductive surgery (mid vaccination, week 12)
  Intratumoral visualization of CD25+ T cells by the [18F]FB-IL2 PET-CT imaging, expressed as standardized uptake values, compared to CD25+ T-cell infiltration in matching tumor material

CONTACTS AND LOCATIONS:
Overall Officials: H. W. Nijman, MD/PhD, Principal Investigator — University Medical Center Groningen, UMCG
Locations (1):
- UMCG, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No